CLINICAL TRIAL: NCT04569110
Title: The Bacteriology of Pleural Infection Using Next Generation Sequencing: The Oxford Pleural Infection Metagenomics Studies (TORPIDS)
Brief Title: The Microbiology of Pleural Infection
Acronym: TORPIDS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 248005
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Pleural Infection; Pleural Infection Bacterial
Keywords: pleural; pleural infection; pleural effusion; microbiome; metagenomics
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Pleural fluid specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pleural infection: Patients with clinically confirmed ongoing pleural infection.
  Interventions: Other: Not applicable. Observational study. Retrospective analysis of samples.
- Negative control: Patients without pleural infection.
  Interventions: Other: Not applicable. Observational study. Retrospective analysis of samples.

INTERVENTIONS:
Other: Not applicable. Observational study. Retrospective analysis of samples. — Not applicable. Observational study. Retrospective analysis of samples.

SUMMARY:
Pleural Infection (PI) is a common, severe and complicated disease with considerable morbidity and mortality. (1,2) The knowledge of pleural infection microbiology remains incomplete. Sequencing of the bacterial 16S rRNA gene is a reliable methodology to discover the total microbiome of complex samples.

The investigators designed a translational metagenomics study to study the bacteriology of pleural infection. The investigators will use pleural fluid specimens from a) the "Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study" (3) clinical trial and b) non-pleural infection patients. The pleural fluid specimens will be subjected to 16S rRNA next generation sequencing.

DETAILED DESCRIPTION:
Pleural Infection (PI) is a common, severe and complicated disease with considerable morbidity and mortality1,2. Patients develop pleural effusions of frankly infected fluid. The understanding of pleural infection microbiome could improve patient clinical management, however the knowledge remains incomplete. Sequencing of the bacterial 16S rRNA gene is a reliable methodology to discovery the total microbiome of complex samples.

The investigators designed a translational study to study the bacteriology of pleural infection. Pleural fluid specimens from a) the "Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study" (3) clinical trial and b) non-pleural infection patients will be subjected to bacterial DNA extraction followed by 16S rRNA next generation sequencing. Moreover, the investigators will study the association between bacterial patterns and important clinical outcomes including survival, duration of hospitalisation and need for surgery.

ELIGIBILITY:
The pleural fluid specimens were collected for the "Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study". PMID: 32675200 DOI: 10.1183/13993003.00130-2020. The investigators analysed the samples retrospectively.

Inclusion Criteria:

* As per protocol of the "Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study". PMID: 32675200 DOI: 10.1183/13993003.00130-2020

Exclusion Criteria:

* As per protocol of the "Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study". PMID: 32675200 DOI: 10.1183/13993003.00130-2020

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with pleural infection (PILOT cohort)
  * Patients with pleural effusion but without pleural infection (negative control group)
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Microbiome | Enrolement
  Discover the microbiome of each sample

SECONDARY OUTCOMES:
Association between bacterial patterns and clinical outcomes | 12 months for survival and requirement for surgical drainage
  Study the association between the microbiome and clinical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Pleural Translational Research, Nuffield Department of Medicine, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies HE, Davies RJ, Davies CW; BTS Pleural Disease Guideline Group. Management of pleural infection in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii41-53. doi: 10.1136/thx.2010.137000. No abstract available. PMID 20696693
- [Background] Corcoran JP, Wrightson JM, Belcher E, DeCamp MM, Feller-Kopman D, Rahman NM. Pleural infection: past, present, and future directions. Lancet Respir Med. 2015 Jul;3(7):563-77. doi: 10.1016/S2213-2600(15)00185-X. PMID 26170076
- [Background] Corcoran JP, Psallidas I, Gerry S, Piccolo F, Koegelenberg CF, Saba T, Daneshvar C, Fairbairn I, Heinink R, West A, Stanton AE, Holme J, Kastelik JA, Steer H, Downer NJ, Haris M, Baker EH, Everett CF, Pepperell J, Bewick T, Yarmus L, Maldonado F, Khan B, Hart-Thomas A, Hands G, Warwick G, De Fonseka D, Hassan M, Munavvar M, Guhan A, Shahidi M, Pogson Z, Dowson L, Popowicz ND, Saba J, Ward NR, Hallifax RJ, Dobson M, Shaw R, Hedley EL, Sabia A, Robinson B, Collins GS, Davies HE, Yu LM, Miller RF, Maskell NA, Rahman NM. Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study. Eur Respir J. 2020 Nov 26;56(5):2000130. doi: 10.1183/13993003.00130-2020. Print 2020 Nov. PMID 32675200